CLINICAL TRIAL: NCT07328217
Title: A Phase 1/2, Open-label, Multicenter Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Antitumor Efficacy of GW5282 in Participants With Advanced Solid Tumors (BEI-DOU2)
Brief Title: A Phase 1/2 Study of GW5282 in Participants With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Dizal Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GW2025EZ0001
Record Dates: First submitted 2025-12-26; First posted 2026-01-09 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2025-12

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dose Escalation Phase (Experimental): Escalating doses of GW5282 administered orally
  Interventions: Drug: GW5282
- Dose Expansion phase (Experimental): The recommended dose(s) for expansion (RDFE) for GW5282 from dose escalation phase will be evaluated in selected tumors.
  Interventions: Drug: GW5282

INTERVENTIONS:
Drug: GW5282 — Single dose period (only for dose escalation phase): administered one single dose at assigned dose level orally.
  Repeated does period (for dose escalation phase and dose expansion phase): administered at assigned dose levels and schedules twice daily (BID) orally in 21-day cycles continuously.
  Arms: Dose Escalation Phase
Drug: GW5282 — RDFE will be determined by dose escalation phase.
  Arms: Dose Expansion phase

SUMMARY:
This is a phase 1/2, open-label, multicenter study assessing the safety, tolerability, pharmacokinetics and efficacy of GW5282 in participants with locally advanced or metastatic solid tumors. This study comprised of a dose escalation phase to determine the MTD and the RP2D and a dose expansion phase to further explore the safety, PK and efficacy of GW5282.

ELIGIBILITY:
Inclusion Criteria:

1. All participants must provide a signed, dated written informed consent (ICF) prior to any study-specific procedures, sampling, and analysis.
2. Male and female participants must be ≥18 years of age at the time of signing the ICF.
3. Eastern Cooperative Oncology Group performance status of 0-1.
4. Histologically or cytologically confirmed locally advanced or metastatic solid tumors who has failed standard of cares (SoCs).
5. Life expectancy ≥3 months.
6. At least one measurable lesion according to RECIST 1.1.
7. Tumor tissue sample requirements: sections of formalin-fixed paraffin-embedded (FFPE) tissue from freshly obtained biopsy sample or archived tumor sample.
8. Adequate organ and marrow function.
9. Participants should be able to comply with the requirements of this study for medication use and follow-up.
10. If the female partner of a male participant has a potential for pregnancy, he must agree to use contraception (such as condoms) and refrain from donating sperm during the treatment period and for at least 6 months after the last dose of study treatment.
11. Female participants should use adequate contraception during the treatment period and for at least 3 months after the last dose of study treatment. Female participants with potential pregnancy should have a negative pregnancy test prior to the first administration of investigational drug. Female participants may also be enrolled if they meet one of the following criteria:

    * Postmenopausal women: older than 50 years and more than 12 months postmenopausal after discontinuation of all exogenous hormone therapy. Women under 50 years of age, more than 12 months postmenopausal after discontinuation of all exogenous hormone therapy, and with luteinizing hormone and follicle-stimulating hormone levels at postmenopausal levels.
    * History of irreversible hysterectomy, bilateral oophorectomy, or bilateral salpingectomy (excluding tubal ligation)."

Exclusion Criteria:

1. Any unresolved > grade 1 (according to CTCAE version 5.0) adverse event (excluding alopecia, anemia, neutropenia, and thrombocytopenia) prior to the first administration of investigational drug.
2. Any known active central nervous system metastases and/or carcinomatous meningitis and/or spinal cord compression.
3. Having any of the following treatment history:

   * previously treated with GW5282 or other EZH pathway inhibitors.
   * previously received any cytotoxic chemotherapy, investigational drug, or other anticancer drug (excluding macromolecular drugs) or clinical trial within 7 days or 5 half-lives (whichever is longer) prior to the first administration of the investigational drug.
   * previously received any macromolecular drug (such as immunotherapy, monoclonal antibodies, bispecific antibodies, or antibody-drug conjugates) within 28 days prior to the first administration of the investigational drug.
   * Underwent major surgery (excluding vascular access surgery) or suffered severe trauma within 4 weeks prior to the first administration of the investigational drug.
   * Received limited field of radiation to alleviate symptoms within 7 days prior to the first administration of the investigational drug, or received more than 30% or extensive field of radiation to the bone marrow within 28 days prior to the first administration of the investigational drug.
   * Received live-attenuated vaccine or viral vector vaccine within 4 weeks prior to the first administration of the investigational drug."
4. Active infectious diseases.
5. History of stroke or intracranial hemorrhage within 6 months prior to the first administration of the investigational drug.
6. History of interstitial lung disease (ILD), radiation pneumonitis requiring corticosteroid therapy, or any clinically active interstitial lung disease, or immunotherapy-related pneumonitis.
7. Uncontrolled systemic disease including uncontrolled hypertension and active bleeding after investigator's assessment.
8. Judgment by the investigator that the participant is unlikely to comply with the study procedures, restrictions, and requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 203 (Estimated)
Dates: Start 2026-01-29 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of Dose Limiting Toxicities (DLTs) (Dose Escalation only) | Up to 21 days
Number of participants with Adverse Events (AEs) | Approximately 24 months from first participant enrolled
Number of Participants with Serious Adverse Events (SAEs) | Approximately 24 months from first participant enrolled
Overall Response Rate (ORR) | Approximately 24 months from first participant enrolled
  ORR is defined as the percentage of subjects with Best Response of Complete Response (CR) or Partial Response (PR) as determined by the investigator

SECONDARY OUTCOMES:
Cmax; Maximum Plasma Concentration of GW5282 | Single dose period (only for dose escalation phase): 0 (predose) up to 72 hours post-dose
AUC; Area Under the Plasma Concentration-time Curve of GW5282 | Single dose period (only for dose escalation phase): 0 (predose) up to 72 hours post-dose
Tmax; Time to Reach Maximum Plasma Concentration (Cmax) of GW5282 | Single dose period (only for dose escalation phase): 0 (predose) up to 72 hours post-dose
Css,max; Maximum Steady State Plasma Concentration of GW5282 | Cycle 1 Day 15: 0 (predose) up to 12 hours post-dose
AUCss; Area Under the Plasma Concentration-time Curve Over the Dosing Interval at Steady State of GW5282 | Cycle 1 Day 15: 0 (predose) up to 12 hours post-dose
Tss,max; Time to Reach Maximum Plasma Concentration (Cmax) at Steady State of GW5282 | Cycle 1 Day 15: 0 (predose) up to 12 hours post-dose
Duration of response (DOR) | Approximately 24 months from first participant enrolled
  DOR is defined as the time from the date of first documented response until date of documented progression, for subjects who achieve CR or PR
Disease Control Rate (DCR) | Approximately 24 months from first participant enrolled
  DCR is defined as the percentage of subjects who have a best overall response of CR or PR or SD as determined by the investigator
Progression-free survival (PFS) | Approximately 24 months from first participant enrolled
  PFS is defined as the time from date of first dose until progression as assessed by the investigator or death due to any cause

CONTACTS AND LOCATIONS:
Overall Officials: Mengzhao Wang, Principal Investigator — Peking Union Medical College Hospital
Locations (3):
- China (3):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Beijing Chest Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality